CLINICAL TRIAL: NCT02337179
Title: A Pilot Study to Introduce Male Circumcision (MC) Services to Prevent HIV Infection in Two High Prevalence Areas of the Dominican Republic (DR)
Brief Title: Male Circumcision Services for HIV Prevention in the Dominican Republic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Instituto Dermatologico y Cirugia de Piel (Unknown)
Responsible Party: Principal Investigator, Maximo Brito, Associate Professor of Medicine & Vice Chair for Urban Global Health, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0863
Record Dates: First submitted 2015-01-07; First posted 2015-01-13 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Circumcision, Male; HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Voluntary medical male circumcision (Experimental): Eligible men will be circumcised according to protocol
  Interventions: Procedure: Voluntary medical male circumcision

INTERVENTIONS:
Procedure: Voluntary medical male circumcision — Male Circumcision Under Local Anesthesia using the Forceps Guided Method

SUMMARY:
The purpose of this study is to determine the feasibility of introducing voluntary medical male circumcision as a form of HIV prevention in high HIV prevalence areas in the Dominican Republic.

DETAILED DESCRIPTION:
Voluntary Medical Male circumcision (VMMC) is an effective strategy to reduce the risk of HIV acquisition in heterosexual men. Observational data and randomized controlled trails (RCTs) conducted in Africa(1,2,3) suggest that the procedure reduces the risk of HIV acquisition by 50-76% in heterosexual males. VMMC has also been shown to reduce the incidence of other sexually transmitted infections (STI), including herpes simplex virus type 2 (HSV-2) and human papilloma virus (HPV) in men(4), and Chlamydia(5), trichomonas vaginalis (TV), bacterial vaginosis (BV) and HPV in their female partners(6).

The results of the RCT's are generating increased demand for safe and affordable MC services in areas of moderate-to-high HIV prevalence where the MC rates are low. Latin America is a region where circumcision of males is uncommon(7). In the Dominican Republic (DR), which is the focus of this study, a 2007 nationwide household survey found that only 13.7% of men between the ages of 15-59 were circumcised(8).

AIDS is the leading cause of death in the Caribbean basin among adults aged 15-44 years. There are approximately 240,000 people currently living with the disease, most of them residing in the Dominican Republic (DR) and Haiti(9). The prevalence of HIV infection in the DR is approximately 0.8% nationwide(8) but it is higher in selected high-risk populations, such as among people living in the "bateyes", the small towns surrounding sugar cane plantations, where the prevalence is 3.2%(10). In pregnant women seeking prenatal care at the main hospital in the Altagracia province HIV seroprevalence is 4.5 %(11). One of the areas of highest prevalence (1.2%) in the country is Region V of health, which includes the provinces of La Altagracia, El Seibo, Hato Mayor, La Romana and San Pedro de Macorís. Prevalence is also higher in the urban slums of the capital city, Santo Domingo.

The public health impact of introducing MC as a strategy to prevent HIV/STI transmission in areas of high HIV/STI prevalence and low MC rates can be significant. In addition to decreasing the rates of HIV and other STI, the intervention could indirectly help decrease the rates of HPV associated cervical cancer. The study proposed here is to develop, implement, monitor and evaluate pilot MC services in selected sites to assess the acceptability, uptake, safety and demand for these services, and to use these data to develop, in collaboration with the Dominican Ministry of Health (MoH), a proposal to the National Institute of Mental Health (NIMH) for support of operations research concerning the safety, uptake, and efficacy of MC interventions in the DR.

1. Specific Aims:

   Based on the results of numerous observational studies and the three RCTs the World Health Organization (WHO) and the Joint United Nations Programme on HIV/AIDS (UNAIDS) have endorsed VMMC as a biomedical intervention for HIV prevention. As such, countries with a high prevalence of HIV in the population are encouraged to examine the feasibility of offering MC services as part of the portfolio of HIV prevention strategies at a national level. The specific aims for this project are:
   1. To develop culturally appropriate education materials about the benefits of VMMC for clients attending pilot healthcare centers.
   2. To train a core group of providers on proper surgical and counseling techniques to provide comprehensive VMMC services.
   3. To determine the acceptability, uptake and demand for MC services in key areas of high HIV prevalence.

      H1: The acceptability and uptake among high risk men will be around 60%.
   4. To assess the safety and adverse events of performing circumcision in resource constrained settings.

      H2: VMMC will result in a complication rate of less than 2%.
   5. To assess sexual risk behaviors, perceptions of sexual function and sexual pleasure in men before and after VMMC. H3: there will be no differences in risk behaviors, sexual function and pleasure after VMMC.
   6. Estimate point prevalence of most common STI in a subset of circumcised men and preserve a small sample of blood to test future scientific hypothesis and/or newer testing techniques as they become available.
   7. To build collaborations with the MoH and other partners in the DR and at UIC to develop a proposal to NIMH for operational research in the context of larger scale MC service provision.
2. Background and significance:

b.1. Male Circumcision to Prevent HIV Transmission Male circumcision is perhaps one of the oldest surgical procedures performed on humans. The millenary practice of removing the male foreskin has cultural, religious and medical dimensions that have been widely studied. Around the world, the procedure is mostly performed for religious reasons in persons of the Jewish and Muslim faiths. Medical indications for MC include phimosis, paraphimosis and balanitis, among others(12). Early evidence of a relationship between MC and HIV infection came from a number of smaller, mostly observational studies, done in Africa(13). These historical data were validated with the completion of three large RCTs in South Africa, Kenya and Uganda, which have shown an overall decrease of 50-76% in the risk of acquiring HIV infection in circumcised males when compared to controls(1,2,3).

The pathogenesis of the initial infection at the level of the foreskin involves tissue macrophages, cell receptors and a moist, poorly keratinized inner prepuce. The first cellular target of the HIV virion on the human genitalia are the tissue dendritic cells in the lamina propria of the submucosa(14). These cells express surface CD4 receptors and CCR5 co-receptors for which HIV has high affinity. In intact human skin, the dendritic cells are shielded from the outer environment by the relatively thick layer of keratin covering the surface of the epithelia. Tissue studies of the human foreskin have shown that the inner lining of the prepuce, exposed during a penile erection, has a thin keratin layer that is very susceptible to microscopic abrasions and can expose the tissue macrophages making them vulnerable to infection by HIV(15).

b.2. MC for STI prevention: MC is an effective strategy to decrease the risk of infection with HIV and other STI in heterosexual males. A beneficial effect has also been observed in decreasing the risk of STI in females. The RCTs confirmed that VMMC decreases herpes simplex virus type 2 (HSV-2) acquisition by 29%, and HPV prevalence by 34% in men(4). Among female partners of circumcised men, bacterial vaginosis was reduced by 40%, and trichomonas vaginalis infection was reduced by 48%(6). Genital ulcer disease was also reduced among males and their female partners by approximately half(16).

b.3. HIV in the Caribbean and the Dominican Republic: The significant decrease in the rate of HIV acquisition observed among circumcised males who participated in the African RCT is generating an increased demand for safe and affordable VMMC services in areas of high HIV prevalence where the procedure is not routinely performed. Latin America is one of such areas where routine circumcision of males is uncommon(7). In the Dominican Republic, only 13.7% of men between the ages of 15-59 years are circumcised(8). The Caribbean is the region of the world with the highest HIV prevalence outside of sub-Saharan Africa (1.0%)(9). Approximately 240,000 individuals are currently living with the disease. Among the Caribbean countries, the Dominican Republic and Haiti report the highest prevalence in the region. According to data from a recent In the DR, the prevalence of HIV infection is 0.8% nationwide(8), however, the numbers are higher in selected populations and in certain geographic locations.

The Dominican healthcare system is administratively divided in 9 regions, which include the country's 31 provinces. Region 0 of health includes the National District and the provinces of Santo Domingo and Monte Plata. The city of Santo Domingo is the capital and financial center of the DR. It has an estimated population of 2.7 million people spread in an area of about 1,400 KM2. 90% of the population lives in an urban setting in this province(17). The overall prevalence of HIV is around 0.7 % in the entire region but is higher in vulnerable groups such as commercial sex workers (CSW) (3.3%), Men who Have Sex with Men (MSM) (5.9%) and drug users (7.1%)(18).

Regions V and VII report the highest prevalence of HIV in the country, 1.2 % and 1.5% respectively(8). Specific populations within these provinces have rates of HIV considerably higher than the national average. For instance, prevalence is 3.2% in the bateyes, the small communities surrounding sugar cane plantations, where a mixed population of Dominicans and Haitian migrant workers cohabitate. Our team has conducted preliminary studies in the Altagracia Province, part of Region V, since it reports the highest province-specific HIV rates and the lowest circumcision rates in the country. A survey of pregnant women seeking prenatal care at the main hospital in the province found an HIV seroprevalence of 4.5 %11. The prevalence of HIV is 5.2% in CSW, 7.6% in MSM and 8.5 % among drug users(18).

c) Preliminary studies: The parent study for this project is a RCT of VMMC to reduce HIV incidence in Kisumu, Kenya whose principal investigator is Prof. Robert C. Bailey, a co-investigator in the current proposal(3). The main objective of that trial was to assess the effectiveness of VMMC in reducing HIV incidence in young, sexually active men. The protective effect found in an intent-to-treat analysis was 53% and in an as treated analysis adjusting for cross-overs and men found to be HIV seropositive at baseline estimated the protective effect to be 60%. Adverse events related to the surgical procedure were few, just 1.5%. Behavioral disinhibition (risk compensation) on the part of circumcised men was small and not significant.

Drs. Brito and Bailey conducted a feasibility study of healthcare facilities in the Altagracia province in the Dominican Republic during June and July of 2007. A total of 37 healthcare facilities were surveyed. The study found that most facilities lacked appropriate equipment to perform surgical procedures and only four (11%) had a surgical theater. 43 healthcare workers, the majority of them physicians (91%), were interviewed for the study. Only 23 % of the personnel had experience performing MC and a significant number of providers (76%) believed they needed comprehensive training in the procedure prior to starting a MC program. Quantitative and qualitative studies to assess the acceptability of MC among men, women and providers in the Altagracia Province were conducted in 2008. In these studies, 73% of men thought that MC improved hygiene and approximately one third knew that it reduces the risk of penile cancer or STI. Only a small percentage (21%) knew that MC helps prevent HIV infection. When first asked, 29% of participants reported that they would be willing to be circumcised if the procedure was offered to them. However, after an educational session detailing the benefits of the procedure for HIV and STI prevention, the acceptability increased to 67%. Such increment was also observed in previous studies done in Botswana(19) and Thailand(20)where acceptability increased from 61 % to 81% and from 14% to 66%, respectively, after a similar information session. In multivariate analysis, the strongest predictors of men's acceptability of circumcision, before the information session, were Haitian nationality (OR=1.86, 95% CI 1.01-3.41), thinking that circumcision improves hygiene (OR=2.78, 95% CI 1.29-6.0) and not believing that having a circumcision decreases sexual pleasure (OR=2.18, 95% CI 1.20-3.94). These results have been published (21, 22).

We also conducted 13 focus group discussions (FGD), 6 with women and 7 with men, each consisting of 6-10 participants (mean=7.9, SD=1.3). One additional FGD was conducted with six physicians, two males and four females, working in rural clinics around the province. Findings of this qualitative study showed that a significant number of participants might be willing to be circumcised, or agree with circumcision for their partners, to improve hygiene, prevent diseases and treat medical conditions, such as phimosis, which can result in pain during intercourse. These results are consistent with our quantitative study on men's acceptability of MC. Perhaps one of the most important findings of the FGD was the enthusiastic endorsement of MC by women, a fact that has potential implications for the successful implementation of a circumcision program in the country (22).

Overall, our preliminary data suggest that men are willing to be circumcised provided they receive information about the benefits of the procedure. Before recommending the introduction of VMMC services as part of a comprehensive package of HIV and other STI prevention strategies, these findings need to be confirmed by studying the uptake of VMMC among sexually active men in selected clinics that serve clients in high prevalence areas. In addition, there is need to identify potential barriers to offering MC services in high risk communities prior to proposing to implement a large-scale intervention. In order to properly address these concerns, we will conduct a pilot study that will provide the necessary preliminary data to design a proposal to the NIMH to conduct operational research around a large-scale implementation project.

d) Experimental design and methods: d.1. Pilot study design The study will be conducted at two sites: the STI clinic at Instituto Dermatologico and Cirugia de Piel (IDCP) in Santo Domingo and the Clínica de Familia in La Romana, Dominican Republic. These sites have been selected on the basis of: 1) high numbers of male clients at risk for HIV and STI infection in communities served by the clinics; 2) high level of acceptability of MC among men in the communities served by the clinics (bateyes of Altagracia); 3) the availability of service providers willing to be trained; 4) the availability of equipment; and 5) the availability of infrastructure, including a minor surgical theater, sterilization facilities and HIV voluntary counseling and testing (VCT) and STI management.

During the first phase of the study, culturally appropriate educational material will be created in Spanish by the principal investigator and local collaborators. Focus Group Discussions (FGD) and in-depth interviews will be conducted with members of the community to learn the educational needs of the community and to assess their opinions on how to best deliver the information on MC that will be contained in the educational materials.

We plan to conduct the FGD in the communities served by the Instituto Dermatologico and the Clinica de Familia, the two main study sites. The plan is to assemble groups of 6-12 participants from the population living in these communities. Community leaders, health promoters, teachers and primary care physicians will be asked to help identify and invite volunteers from their respective communities to participate in the study. There will be no difference in the recruitment process for men and women. They will be recruited from the same venues (schools, clubs, community centers) . Participants will be invited to participate by research personnel with the help of local leaders. These local leaders may be of both genders and will help recruit participants from either gender. The focus groups will be gender-specific. The moderator will explain the purpose of the study to participants. Verbal consent will be obtained from all participants and an information sheet outlining the objectives of the study, their privacy and confidentiality rights and our contact information will be distributed. The document will highlight the voluntary nature of the subject's participation and their right to leave the discussion at anytime if they so desire. The study meets the definition of "minimal risk", therefore, we are requesting a waiver of written consent. We believe this will further preserve the confidentiality of the participants. The goal is to conduct no more than 15 FGD. Participants in the FGD will be divided by gender. We plan to recruit approximately the same number of men and women for the FGD.

In addition to the FGD, several in-depth individual interviews may be conducted using the same guide than in the FGD. A script will be followed to conduct the FGD. The discussions will be stimulated by using a list of carefully crafted questions on the subject of MC. These questions are designed to obtain information on the following aspects relevant to our investigation:

1. Perception of the population about the frequency of MC in community men.
2. Opinions on the best way to educate men in the community about the benefits of circumcision.
3. Opinions about the content of the educational materials educational and how information should be delivered.
4. Where should these educational material be posted or distributed to capture the most number of men.
5. Opinions on the best venue to organize educational sessions featuring a circumcised man that would be available to answer question from men in the community about his satisfaction with his circumcision.
6. Perceptions about who would be a good person to educate men about the benefits of circumcision in the community.
7. Opinions on the best way to involve women in the community in a campaign to recruit men for circumcision.

The moderator and a research assistant (RA) will lead the discussions. All FGD will be audiotaped and detailed notes will be taken. The content of the recordings will be transcribed shortly after the end of the meeting. The PI, a native Spanish speaker, will be responsible for translating the recordings from Spanish to English. The English-version transcripts will be coded using the program ATLAS.ti vers. 5.2 based on template of topical categories drawn from questions and issues covered in the discussion guides and from themes emerging from the discussions themselves. The interviews will be conducted by one of the co-investigators. Verbal consent will be obtained and a document containing information about the study will be provided to the participants. All data obtained during this study, including recordings and notes will be de-indentified. The names of the participants will not be recorded to protect their confidentiality.

Data Management All notes, audio recordings and study material obtained during the FGD and interviews will be kept in a locked filing cabinet in an office at the Instituto Dermatologico, Dominican Republic and in the PI's office at the UIC campus upon the investigator's return to Chicago. All data will be de-identified to preserve confidentiality. Names will not be recorded. Verbal informed consent will be sought; there will be no signed consent forms to identify individuals. The participants have the right to review the audio recordings. If a participant requests to listen to the recordings, one of the co-investigators will schedule an appointment for the subject to come to the research site and, in an unoccupied office, will playback the recording for him/her and answer all the questions that the subject may have. If the participant wishes to erase part or all of his/her responses, it will be done on the spot, in his/her presence, using the digital recorder. The data obtained during these FGD and interviews will inform the design of the educational materials. Once created, these materials will be tested for clarity and appropriateness of language by soliciting input from community health promoters and peer advocates working at the IDCP. Once it is determined that the educational materials are suitable to distribute to clients, we will submit to the Institutional Review Board for approval. Once approved, pamphlets and posters will be printed and distributed at the site clinics and the surrounding communities.

During the second phase, selected providers will be trained. This will include counselors in HIV counseling and testing, and medical doctors by an experienced urologist on the appropriate technique for VMMC using the "Manual for Male Circumcision Under Local Anesthesia" published by WHO, UNAIDS. Supervision and evaluation of trainees will be conducted following the protocol used during the parent RCT.

Study subjects will be recruited in a variety of ways. In Santo Domingo, fliers will be posted in bars and night clubs frequented by men at high risk for HIV/STI acquisition. A group of volunteer commercial sex workers working on an HIV vaccine trial will be asked to refer their clients for the study. Men seeking care for STI at the clinic will also be invited to participate. In La Romana, men attending the Clínica de Familia will be invited to participate. In addition, a group of outreach workers will visit the "bateyes", the communities surrounding sugar cane fields where migrant laborers live, to educate men about MC and invite them to participate in the study.

Men between 18-40 years will be provided with information about the study and will be invited to participate. If they express an interest in participating, informed consent will be obtained. The participant will go over the consent form with the counselor, who will assess his level of understanding and answer any questions. If there are no temporary or permanent excluding conditions, the participant will be asked to give informed consent for enrollment in the study. Men who elect to be circumcised will be fully informed about the benefits and risks of the procedure, as well as the surgical method to be used. After the informed consent is signed, a "Locator Information Form" containing confidential data such as subject's name and address will be completed. Only selected research staff will have access to this information, which will be filed separate from the rest of the study forms. A de-identified "demographic information form and behavioral questionnaire" will be completed next.

Testing for HIV infection will be carried out using a rapid test. The test kits to be used are the synthetic peptide test, Determine HIV 1/2, and the recombinant antigen test Unigold HIV 1/2 Recombinant. Results are provided to the clients, with appropriate counseling, at the same visit. Participants are taught to observe, read and interpret the tests for themselves in the company of the counselor. Men with positive results will be informed of their HIV status and will be followed-up at the study clinic and referred for a confirmatory HIV-ELISA and, if confirmed, for HIV treatment. Serologic testing for HSV-2, hepatitis B surface antigen (HBV), and hepatitis C antibody (HCV) will be performed using an ELISA test. A serum Rapid Plasma Reagin test (RPR) will be performed to test for syphilis. Chlamydia and gonorrhea testing will be performed in urine using a Polymerase Chain Reaction (PCR) assay. All participants who test positive for Chlamydia, syphilis and gonorrhea will be offered treatment free of charge. Participants who test positive for HSV-2 and have active genital lesions will be offered treatment free of charge. Those who test positive but have no active lesions will be counseled on safe sex practices and the risk of transmission to their partners as there is no recommended treatment for asymptomatic individuals infected with HSV-2. HIV, HBV, and HCV positive participants will be referred for evaluation and treatment at Clinica de la Familia in La Romana as these are chronic diseases that require long term treatment usually covered under government programs. If a participant is found to have a treatable STD and he does not return to the site, he will be called by the study investigators using the phone number provided by the participant at enrolment to ensure treatment is provided. If there is a temporary, medically curable condition present, such that it would be advisable to defer potential surgery, then the participant will be treated and asked to return for re-evaluation for study eligibility when he is cured. Men found to have an STD or to be HIV-positive will be referred for immediate care. Once enrollment is completed, participants will be given an appointment for the surgery.

Circumcision will be performed soon after informed consent, preferably within a few days. All surgeries will be done under local anesthesia in a clinic by trained clinicians, using the standardized forceps-guided method described by Krieger and colleagues and contained in the WHO MC manual(23). Circumcised men will be counseled to refrain from sex for six weeks post-surgery and counseled about risk of HIV infection through open wounds during the healing process. They will be checked for complications and asked about their sexual activity seven days after the procedure. Men without complications will be followed six months after surgery with behavioral risk assessment, HIV testing and counseling. Men may come to the study sites for unscheduled visits at any time during the 6 month follow-up. All men will be counseled at enrollment and all follow-up visits to reduce their risk for HIV infection by consistent condom use and, where applicable, reductions in numbers of sex partners. Counselling on condom use and sexual risk reduction will be provided by trained, experienced, native-speaking counsellors.

MC services will be offered at the selected two sites for 1 year. The estimated cost per circumcision is $40. We expect to recruit five clients per week at each site for a total convenience sample of 575 subjects in one year. During the second year of the project, we will continue to assess behavioral risk factors for the first six months and work on analyzing the data during the last semester of the project.

Circumcision Procedure Prior to surgery, the clinician will obtain a complete medical history and perform a physical exam.

A brief description of the procedure follows. The patient lies on his back in a comfortable position. The pubic area is shaved clean with a disposable razor and the hair is picked up with a dressing tape. The surgeon scrubs up and puts on 2 pairs of sterile gloves. The client's skin is prepared with Betadine solution, making sure that the inner surface of the prepuce and the glans are clean and the skin is dry. The outer pair of gloves is then removed. The client is draped with two drapes and a center "O" towel, and then, using 2% lidocaine without epinephrine, a dorsal nerve block and a field block with special attention to the ventral nerve, is performed. Normally, no more than 10ml of 2% lidocaine will be used. The anesthetic effect of the nerve block is checked, and revised if necessary. The prepuce is held with two mosquito forceps, one on each lateral aspect, then a curved mark is made with sterile disposable marking pens, outlining the planned surgical cut. The mark is made one cm proximal to the coronal sulcus all round, and parallel to the coronal sulcus. The prepuce is clamped along the mark with a Kocher clamp while retracting the glans, ensuring that the glans itself is not clamped. The prepuce is excised using a surgical blade along the mark. Bleeders are identified, clamped and tied. They are sutured, and if necessary ligated, using 3/0 plain catgut. After ligating all the bleeders, the area is irrigated with normal saline and then inspected for more bleeders, which are identified and tied. Using 3/0 chromic catgut on a taper 4/8 circle needle, a U-shaped horizontal mattress stitch is made on the ventral side of the penis (frenulum) to join the skin at the "V" shaped cut, which is then tied and tagged with a mosquito forceps. Using vertical mattress stitches, four quarters are tagged, and a vertical mattress stitch added, after which a simple stitch is put at the center of every two mattress stitches (a total of at least 16 stitches). The area is irrigated with normal saline and other simple stitches added as required. The wound is dressed with Sofratulle, then with a regular dressing bandage and a strapping. The client is advised to rest for 30 minutes, and if stable, discharged home on mild analgesics. Upon completion of the procedure the surgeon completes a procedure form. The excised foreskin tissue is taken to the laboratory with no identifiers, discarded with other laboratory waste, and incinerated with other biological waste within three days. Participants will be given verbal and written instructions on postoperative wound care and counseled to refrain from sexual activity for at least six weeks after the procedure. They will also be encouraged to come to the clinic or contact a clinician at any time with medical problems.

Day 7 Post Circumcision Visit: Circumcised men will be asked to return to the clinic 7 days after the procedure to check the wound, to see if it is healing properly, to check for complications, and to ask about their sexual activity, their level of pain, resumption of work or other activities, and their satisfaction with the procedure and care at the clinic. As with all visits, any adverse events will be recorded. Blood and urine will be collected for STD testing at this visit.

Six month post operative visit: During this visit a brief exam to confirmed proper wound healing will be performed. A behavioral and satisfaction questionnaire will be administered.

Unscheduled Follow-up Visits: Ad hoc clinic visits will be encouraged to check and treat for complications of the procedure. At such visits, medical examinations and laboratory testing will be conducted as indicated, and appropriate treatment provided free of charge. Medical referral will be made if required.

d.2. Data analysis Each enrolled participant will be assigned a confidential code, which will be used in all study forms. Only the principal investigators and research assistants will have access to the "locator information form" containing personal information. This form, which links the subject's confidential code to his name, will be stored in separate locked filing cabinets at the local principal investigator's offices. The locator information forms, which contain the personal information on the subjects, will be kept for 1.5 years in case we need to contact one of the subjects for an unexpected occurrence or with a question. After the end of that period, these locator forms will be destroyed at the research offices at the respective study sites using a micro cut shredder. Data will be coded and entered into computer datasets by trained personnel. Data extracted from questionnaires will be tabulated and analyzed using SAS statistical software version 9.1. and will be analyzed at the University of Illinois, College of Medicine, in Chicago by the principal investigator A questionnaire asking specific demographic information will be administered. The following variables will be recorded: age, religion, place of residence (urban/rural), education level, occupation and marital status. Simple descriptive statistics will be calculated and the effect of these variables on the willingness, uptake and rate of adverse events of VMMC will be estimated. In addition, we plan to estimate the effect of demographic characteristics on sexual behavior and disinhibition after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Uncircumcised men;
2. Aged 18-40 years

Exclusion Criteria:

1. Foreskin covering less than half of the glans;
2. Bleeding disorders;
3. Keloid formation;
4. Other conditions that might unduly increase the risks of elective surgery.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 539 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants who agreed to undergo circumcision after being offered. | 13 months

SECONDARY OUTCOMES:
Number and percentage of adverse events by severity (mild, moderate, severe) | 23 months
Number and percentage of individuals who use illicit drugs | 23 months
Number and percentage of men who have sex with men | 23 months
Number and percentage of individuals who had ≥ 2 sex partners over the last 30 days | 23 months
Number and percentage of individuals who experienced problems with penis and foreskin prior to circumcision | 23 months

CONTACTS AND LOCATIONS:
Overall Officials: Maximo O Brito, MD, MPH, Principal Investigator — University of Illinois at Chicago; Yeycy Donastorg, MD, Study Director — Instituto Dermatologico y Cirugia de Piel
Locations (2):
- University of Illinois at Chicago, Chicago, Illinois, United States
- Instituto Dermatologico y Cirugia de Piel, Santo Domingo, Dominican Republic

REFERENCES:
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] Tobian AA, Serwadda D, Quinn TC, Kigozi G, Gravitt PE, Laeyendecker O, Charvat B, Ssempijja V, Riedesel M, Oliver AE, Nowak RG, Moulton LH, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH. Male circumcision for the prevention of HSV-2 and HPV infections and syphilis. N Engl J Med. 2009 Mar 26;360(13):1298-309. doi: 10.1056/NEJMoa0802556. PMID 19321868
- [Background] Castellsague X, Peeling RW, Franceschi S, de Sanjose S, Smith JS, Albero G, Diaz M, Herrero R, Munoz N, Bosch FX; IARC Multicenter Cervical Cancer Study Group. Chlamydia trachomatis infection in female partners of circumcised and uncircumcised adult men. Am J Epidemiol. 2005 Nov 1;162(9):907-16. doi: 10.1093/aje/kwi284. Epub 2005 Sep 21. PMID 16177149
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Nalugoda F, Watya S, Moulton L, Chen MZ, Sewankambo NK, Kiwanuka N, Sempijja V, Lutalo T, Kagayii J, Wabwire-Mangen F, Ridzon R, Bacon M, Wawer MJ. The effects of male circumcision on female partners' genital tract symptoms and vaginal infections in a randomized trial in Rakai, Uganda. Am J Obstet Gynecol. 2009 Jan;200(1):42.e1-7. doi: 10.1016/j.ajog.2008.07.069. Epub 2008 Oct 30. PMID 18976733
- [Background] Drain PK, Halperin DT, Hughes JP, Klausner JD, Bailey RC. Male circumcision, religion, and infectious diseases: an ecologic analysis of 118 developing countries. BMC Infect Dis. 2006 Nov 30;6:172. doi: 10.1186/1471-2334-6-172. PMID 17137513
- [Background] CESDEM. Encuesta Demográfica y de Salud, República Dominicana. 2007. (accessed January 2, 2010 at (http://www.cesdem.com/html/encuesta_demografica_y_de_salud_2007.pdf )
- [Background] Joint United Nations Programme on HIV /AIDS. 2009 Report on the global AIDS epidemic. (Accessed February 2, 2010 , at http://www.unaids.org/en/KnowledgeCentre/HIVData/GlobalReport/
- [Background] CESDEM. Encuesta Sociodemográfica y sobre VIH/SIDA en los Bateyes Estatales de la República Dominicana. 2007. (accessed January 2, 2009 at http://www.cesdem.com/html/encuesta_sociodemografica_y_sobre_vih_sida_en_los_bateyes_estatales_de_la_republica_dominicana.pdf )
- [Background] Secretaria de Estado de Salud Publica. Encuesta de seroprevalencia de la infección VIH basadas en puestos centinela. 2006.
- [Background] UNAIDS. Male circumcision: global trends and determinants of prevalence, safety and acceptability. (accessed February 23, 2010 at ( http://whqlibdoc.who.int/publications/2007/9789241596169_eng.pdf )
- [Background] Weiss HA, Quigley MA, Hayes RJ. Male circumcision and risk of HIV infection in sub-Saharan Africa: a systematic review and meta-analysis. AIDS. 2000 Oct 20;14(15):2361-70. doi: 10.1097/00002030-200010200-00018. PMID 11089625
- [Background] Kahn JO, Walker BD. Acute human immunodeficiency virus type 1 infection. N Engl J Med. 1998 Jul 2;339(1):33-9. doi: 10.1056/NEJM199807023390107. No abstract available. PMID 9647878
- [Background] McCoombe SG, Short RV. Potential HIV-1 target cells in the human penis. AIDS. 2006 Jul 13;20(11):1491-5. doi: 10.1097/01.aids.0000237364.11123.98. PMID 16847403
- [Background] Gray RH, Serwadda D, Tobian AA, Chen MZ, Makumbi F, Suntoke T, Kigozi G, Nalugoda F, Iga B, Quinn TC, Moulton LH, Laeyendecker O, Reynolds SJ, Kong X, Wawer MJ. Effects of genital ulcer disease and herpes simplex virus type 2 on the efficacy of male circumcision for HIV prevention: Analyses from the Rakai trials. PLoS Med. 2009 Nov;6(11):e1000187. doi: 10.1371/journal.pmed.1000187. Epub 2009 Nov 24. PMID 19936044
- [Background] ONE. VIII Censo nacional de poblacion y vivienda 2002. (accessed February 23, 2010 at(http://onedatabase.indotel.net.do/cgibin/RpWebEngine.exe/PortalAction?&MODE=MAIN&BASE=CPV2002&MAIN=WebServerMain.inl )
- [Background] COPRESIDA. Primera encuesta de vigilancia de comportamiento con vinculacion serologica en poblaciones vulnerables 2008. 1: 39-88.
- [Background] Kebaabetswe P, Lockman S, Mogwe S, Mandevu R, Thior I, Essex M, Shapiro RL. Male circumcision: an acceptable strategy for HIV prevention in Botswana. Sex Transm Infect. 2003 Jun;79(3):214-9. doi: 10.1136/sti.79.3.214. PMID 12794204
- [Background] Tieu HV, Phanuphak N, Ananworanich J, Vatanparast R, Jadwattanakul T, Pharachetsakul N, Mingkwanrungrueng P, Buajoom R, Teeratakulpisarn S, Teeratakulpisarn N, Methajittiphun P, Hammer SM, Ann Chiasson M, Phanuphak P. Acceptability of male circumcision for the prevention of HIV among high-risk heterosexual men in Thailand. Sex Transm Dis. 2010 Jun;37(6):352-5. doi: 10.1097/OLQ.0b013e3181c9963a. PMID 20145588
- [Background] Brito MO, Caso LM, Balbuena H, Bailey RC. Acceptability of male circumcision for the prevention of HIV/AIDS in the Dominican Republic. PLoS One. 2009 Nov 2;4(11):e7687. doi: 10.1371/journal.pone.0007687. PMID 19888322
- [Background] Brito M, Luna M, Bailey RC. Feasibility of introducing male circumcision (MC) in the Dominican Republic : AIDS 2008 - XVII International AIDS Conference: Abstract no. MOPE0548.
- [Background] WHO. Manual for MC under local anesthesia 2009. (accessed February 23, 2010 at(http://www.who.int/hiv/pub/malecircumcision/local_anaesthesia/en/index.html )
- [Derived] Brito MO, Lerebours L, Volquez C, Basora E, Khosla S, Lantigua F, Flete R, Rosario R, Rodriguez LA, Fernandez M, Donastorg Y, Bailey RC. A Clinical Trial to Introduce Voluntary Medical Male Circumcision for HIV Prevention in Areas of High Prevalence in the Dominican Republic. PLoS One. 2015 Sep 14;10(9):e0137376. doi: 10.1371/journal.pone.0137376. eCollection 2015. PMID 26367187